CLINICAL TRIAL: NCT03663322
Title: Diabetes and Osteopathic Manipulative Medicine: A Randomized Controlled Trial
Brief Title: Diabetes and Osteopathic Manipulative Medicine (OMM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Institute of Technology (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BHS-1383
Record Dates: First submitted 2018-09-05; First posted 2018-09-10 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Type2 Diabetes Mellitus; Osteopathy in Diseases Classified Elsewhere

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessor will be blinded to the arm the participants have been randomly assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT Protocol (Experimental): Subjects assigned to this arm will have selected osteopathic manipulative treatment techniques administered during the treatment sessions
  Interventions: Procedure: OMT Protocol
- OMT-Sham Protocol (Sham Comparator): Subjects assigned to this arm will have sham-osteopathic manipulative treatment techniques administered during the treatment sessions
  Interventions: Procedure: OMT-Sham Protocol

INTERVENTIONS:
Procedure: OMT Protocol — Selected hands-on OMT techniques intended to improve pancreatic function will be administered during the treatment sessions
  Arms: OMT Protocol
Procedure: OMT-Sham Protocol — Selected hands-on Sham-OMT techniques that are not intended to affect pancreatic function will be administered during the treatment sessions
  Arms: OMT-Sham Protocol

SUMMARY:
Our research team is proposing a study to investigate the effects of osteopathic manipulative treatment on the blood sugar levels of persons with Type 2 diabetes. The goal of this study is to determine if osteopathic manipulative treatment (OMT) can improve the blood sugar levels of individuals with Type 2 diabetes. Half of the participants will receive osteopathic manipulative treatment (OMT) and the other will receive OMT-sham treatment.

DETAILED DESCRIPTION:
The Research Plan

Aims Type II diabetes is a common endocrine disorder of glucose metabolism that is linked to considerable morbidity and mortality. In the United States, diabetes is a major cause of cardiovascular disorders including heart disease and stroke. It continues to rise in prevalence despite the advances made in methods of diabetic glucose control. Diabetes is a complex chronic disease that involves continuous medical care and self-management strategies. The main treatment strategies consist of medications and lifestyle modifications. However, the strategies used in clinical trials while effective are impractical as they are intensive and expensive to ensure maintaining these treatment strategies over time. A major opportunity exists for treatment modalities that are affordable and readily implementable such as OMT.

Osteopathic literature suggests that there may be a role for OMT in the treatment of patients with diabetes mellitus. This is supported by our preliminary data reported below. The OMT protocol developed for this research study is based on osteopathic literature and geared towards optimizing bodily function for patients with Type II diabetes and blood-glucose homeostasis. OMT utilizes manual forces directed to improve physiological function and homeostasis by reducing localized dysfunctions of the body referred to as somatic dysfunctions. OMT may be beneficial in reducing blood glucose levels in Type 2 diabetic individuals. Improving glucose levels in type II diabetics would reduce the morbidities and complications of this disorder and have a large impact on patients' health outcomes as well as in healthcare systems worldwide.

Specific Aims: To determine if the OMT protocol outlined in this study will improve glucose and A1C levels in individuals with Type II diabetes.

1. To investigate whether the use of OMM (osteopathic manipulative medicine) targeting pancreatic function will decrease blood glucose in diabetic patients after each OMM treatment (short-term effects)
2. To investigate whether the use of OMM targeting pancreatic function over a 3 month period will decrease blood glucose in diabetic patients (long-term effects)
3. To investigate whether the use of OMM targeting pancreatic function over a 3 month period will decrease A1C levels in diabetic patients (long-term effects)

The primary outcome measure for glucose levels will be measured by obtaining pre and post OMT/OMT-sham glucose levels at each of the 6 treatments sessions delivered every 2 weeks for 3 months. The primary outcome measure for A1C levels will be measured by obtaining blood samples at time 0, at the end of months 1, 2 and 3. Results will be compared between the OMT and OMT-sham groups. If the results support the hypotheses, the OMT protocol can be filmed on video and performed in workshops for other osteopathic physicians to improve glucose control in their Type II diabetic patients.

Background A comprehensive systematic review of the published osteopathic literature found little evidence of OMT as part of the management of Type II diabetes. Nevertheless, the few published articles do provide encouragement for future studies on this topic. A small study, which was subsequently re-analyzed, suggested that OMT may reduce blood glucose levels and increase insulin secretion in diabetic patients. In this study 150 diabetic patients had fasting blood glucose measured and this was followed by provision of OMT targeted to produce pancreatic stimulation and glucose levels. The patients had glucose measured either 30 minutes and/or 60 minutes after the OMT session. The results obtained revealed a rapid decrease in the glucose levels of the treated patients. The investigators have obtained similar results during the course of our care of Type II diabetic patients. A case-control pilot study found consistent osteopathic palpatory findings in patients with Type II diabetes as compared to the non-diabetic patients. Other osteopathic literature support the use of OMT in the treatment of diabetes-related musculoskeletal complications In light of the little evidence of previously published osteopathic literature and the potentially high impact that the results would have, the investigators propose to conduct a study to investigate the possible effects of OMT on glucose and A1C levels in patients with diagnosed Type II diabetes as compared with an OMT-sham treatment protocol. The goals of this study will be to determine if OMT is effective in the management of patients with Type II diabetes.

Power analysis/methods:

Power analysis has been performed to estimate an optimal sample size required to achieve at least 80% of statistical power in the ANCOVA analysis. An effect size as a necessary input for power analysis was estimated based on the information in the reference that investigated the effects of an education program with exercise on blood glucose and A1C levels in subjects with Type 2 diabetes. A total of 90 Type II diabetic subjects is required to detect the estimated effect size of d=0.6 with a statistical power of 80% and α=0.05. After accounting for an expected attrition rate of 10%, a total of 100 subjects with Type II diabetes will be recruited.

The trial will be registered on clinicaltrials.gov. Recruitment will be the primary focus in the first 3 months of the study. All of the above manners of recruitment will be re-visited every 3 months until the trial is completed.

Research design and methods Subjects: Participants with diagnosed Type II diabetes will be randomized into the OMT intervention or OMM-sham cohorts for comparison of the effects of the OMT protocol on our outcome measures.

Subject population characteristics:

Sample size: 100 Age range: 30-90 years Gender: Male or female Racial/ethnic background: any Health status: Type II diabetic diagnosed at least 5 years prior to inclusion in this study

Specimens, records, and data: will be collected from individual participants in this study. Blood glucose and A1C levels will be obtained using a Glucometer and A1C kits and will be processed and recorded at the time of the visit.

Recruitment Plan:

Subjects will be recruited by direct recruitment from the NYIT Academic Health Care Center and Family Health Care centers, posting of IRB-approved flyers in local public places, contact with local endocrinologists to identify interested patients and introduce the study at local Diabetic disease support groups and symposiums. The NYIT Academic Health Care Center and Family Health Care Centers in which the investigators see patients provides healthcare services to over 500 patients with Type II diabetes annually. The investigators will directly recruit participants for this clinical trial using these recommendations. IRB-approved flyers will be placed in visible areas of our health centers. The flyer will have the principal investigators name, office number, and email address for potential participants. The organizers for local support groups and symposiums for Diabetes will be contacted. The principal investigator will request to attend the meeting to provide a brief introduction to the study and recruit participants that may meet the eligibility criteria. Other local endocrinologists may be called to introduce the study and to request that these specialists identify any of his/her patients that may be interested in our research.

Consent procedure:

Recruited, eligible subjects will be presented with the consent form and given as much time to read or have the form read to them as necessary to decide. A faculty investigator will be present during this process to answer any questions the subject may have. The consent to their participation in the study using a written form will be obtained by a faculty investigator.

Potential risks to participants:

Subject may experience minor emotional distress from talking about their medical history or the structural physical exam. As with all individuals treated with OMT, the subject may experience soreness after the OMT. The subject may experience discomfort from the blood glucose testing. The risks associated with fingersticks for the blood glucose and A1C levels include risk of bleeding, infection, or syncope. Standard precautions during fingerstick procedures will be followed. Alternatively, subjects may benefit by becoming more aware of various aspects of their diagnosis.

Protection against risks:

In the case of any adverse effect from this study, Sonia Rivera-Martinez, DO, Karen Sheflin, DO or Jayme Mancini, DO, PhD, will be contacted about the incident and the subject will cease any participation in the research study. In addition, the Institutional Review Board (IRB) will be notified of the adverse effect within 24 business hours. No deception will be used in this study. If the research should reveal a medical or potentially troubling condition, the subject will be advised to make an appointment with their primary care physician. Semi-annual progress reports and annual renewal reports to the NYIT IRB are required for all IRB-approved protocols. Any adverse effects will be evaluated by the full IRB. Note that this research protocol will be submitted for IRB approval.

Participation in the study will be entirely voluntary and confidential. In the study, the subjects will be given a number for blinding purposes. Each subject will be assigned and given a registration identification that does not contain any content that can identify the subject. For example, IRB1130_PDC001 will be the subject identification for the first subject and IRB1130_PDC002 will be for the second subject and so forth. The subject's name, date of birth or other identifying material will not be included in this file. The subject's number identity will be secured in the office of the principal investigator on a desktop computer requiring a login and password for access.

Access to the subject's information will be allowed only by the research team to ensure confidentiality. The questionnaire and test data will not have patient identification information and if it is printed out and it will be stored under lock and key in the principal investigator's office. If it is not printed out, it will be kept on a password protected on our computer. Since there is no identifying material for each subject file only the investigators will know which data correlates with which subject. Thus, subject data is safeguarded in a HIPAA compliant program and is separated from any clinical patient files. The process of maintaining human research subject confidentiality is practiced by NYITCOM faculty, staff, and students and monitored by the Assistant Dean of Research and the NYIT IRB.

Risks to subjects:

The methods utilized in this study are minimal risk and not different than are used in standard health care. There may or may not be a direct benefit to the subjects during the study, however, the information taken from the study may benefit the subjects or other people with Type II diabetes in the future.

Outcome Measures (A) Fasting glucose levels: Each participant will be tested 12 times throughout the course of their individual participation in the research study. The fasting glucose levels will be obtained pre-OMT/OMT-sham and 30 minutes post-OMT/OMT-sham treatments have been completed. Each OMT/OMT-sham session will last 15 minutes and will be scheduled from (8 AM to 10 AM). Each participant will have a total of 6 treatment sessions which will be scheduled every 2 weeks. Specific glucometer test kits will be utilized for the purpose of obtaining the glucose levels. The subjects will be scheduled for the OMT/OMT-sham treatments at the same time slot for each visit to decrease the likelihood of glucose variability due to the measurements being taken at different times of the day. (Refer to Appendix A - Protocol for fasting glucose)

(B) A1C levels: Each participant will be tested 4 times throughout the course of their individual participation in the research study. The A1C levels will be obtained pre-OMT/OMT-sham at their 1st visit and at the end of their 2nd, 4th and 6th visits. A1C levels have an approximate ½ life of 28 days. It is, therefore, reasonable to expect a change at around this timeframe.

All participants will be scheduled for their first visit, which will include documentation of meeting eligibility criteria, consenting, and assignment to a cohort, first visit outcome measures, and first OMT or OMT-sham as assigned. The primary outcome measures of glucose levels will be assessed at pre and post OMT/OMT-sham at each of their 6 visits which will be scheduled every 2 weeks for 3 months.

Subjects will be instructed to maintain the same physical activity level, continue their current diet and avoid changes in these throughout the trial period. Should any change occur subjects will be advised to inform one of the study investigators. This last is to decrease the likelihood of variations in glucose levels due to changes in physical activity levels or dietary changes.

OMT Protocol for Type II Diabetes: Weeks 1-6:

Previous reports suggest that primary areas of the body particularly important for blood-glucose homeostasis include the autonomic nervous system (parasympathetic innervation via the vagus nerve, sympathetic innervation of the pancreas and liver and kidneys and adrenal glands), thoracolumbar diaphragm, abdominal lymphatic system (including mesentery), and the pancreas, liver, and adrenal glands themselves.

The investigators have selected techniques for the OMT protocol which were used by Dr. Bandeen in his study in which glucose levels were reduced and those recommended in other studies for the treatment of Type 2 diabetes. Refer to list below.

1. Suboccipital release
2. Thoracic outlet release
3. Rib raising Left ribs 2-9 right ribs 5-12 and ribless rib raising right L1-2
4. Chapman's points for pancreas and liver
5. Fascial Stretch of the Pancreas in Longitudinal Axis
6. Test and Treatment of Pancreatic Motility
7. Pancreatic Fascial Technique
8. Pancreatic stimulation through angle of ribs 3-5
9. Celiac ganglion inhibition
10. Liver pump

The above techniques are well described in the osteopathic literature. The OMT-Sham protocol will involve simply placing the hands in the general areas of where the OMT selected OMM techniques are administered. Each technique will be performed for approximately one minute each.

All treating physicians will have Board certification by the American Osteopathic Association (AOA) to perform Osteopathic Manipulative Treatments. There will be 2 physicians who will be specifically trained to deliver either the OMT or OMT-Sham treatment protocols. This measure will ensure that the techniques are performed in a uniform manner. Every physician will treat an approximately equal number of subjects.

The treating physicians will be instructed to execute the OMT and OMT-Sham treatment techniques in the exact order as listed and described in this proposal. The manipulative techniques of the OMT protocol are those that have been well described in standard osteopathic textbooks. The sham treatment protocol for this study was designed to be analogous to the OMT regimen with respect to the treatment time, areas treated and positioning of the subjects.

Expectations for the proposed study:

If the OMT protocol is effective in treating Type II diabetic subjects the investigators expect a reduction in the glucose levels in the short term and long term and a reduction in the A1C levels over the course of the research study.

Analysis To investigate the primary specific aims, analysis of covariance (ANCOVA) will be used to compare the changes in the before and after treatment sessions for the OMT and OMT-sham groups with a statistical power of 80% and α=0.05. Analyses will be conducted using IBM SPSS Statistics 22.

Potential difficulties and limitations of the proposed procedures and alternative approaches to testing the hypotheses:

Difficulties associated with this study have been addressed where possible. Variability in the Type II diabetes histories and their associated symptoms will be addressed by analyzing their effects on the outcome measures. The high attrition rate associated with the diabetic participants is addressed by planning to recruit an extra 10% of the expected number needed for significance. There may be a sampling bias wherein people with Type II diabetes and may be more likely to pursue treatments at our health centers due to the variety of providers available and social support.

Time-table The OMT protocol was developed by utilizing the available osteopathic literature and the testing of the administration of the protocol by PI's on her Type II diabetic patients. Testing the OMT protocol to prove significant improvements in glucose and A1C levels function amongst individuals with Type II diabetes in a randomized controlled trial is necessary. Recruitment efforts will continue until the sample size required for significance is reached as described in the analysis. Statistical analysis will be calculated every 6 months to determine trends in primary outcome measures and assess any reported side effects. If risks out-weigh benefits, consider modification of methods or termination. The final statistical analysis will be done at the completion of the trial.

APPENDIX A - Protocol for Fasting Glucose

Instructions to subjects for fasting blood glucose:

* Do not eat or drink anything but water for eight hours before the appointment in which the fasting blood glucose measurement will be taken.
* Hold off from taking their diabetes medications until after the research encounter has been completed.
* Please report immediately to the investigator taking the fasting blood glucose measurement if the participant has or feels any of the following symptoms at any time during the research encounter:

  * Sweatiness and shakiness
  * Weakness
  * Confusion
  * Irritability
  * Pale
  * Rapid heart rate
  * Uncoordinated
  * Excessive fatigue
  * Blurry vision

Instructions for research staff, investigators, and physician investigators:

Subject with hypoglycemia: Fasting blood glucose < 70 and/or with any of the above symptoms:

1. Provide patient with a small glass of orange or apple juice or Glucerna shake. Contact a physician investigator to evaluate the subject. Physician investigator will make the clinical decision if the patient should be referred to the nearest emergency department or can be safely discharged to their home.
2. The patient will not have OMT/OMT-sham treatment given at that specific research encounter

Subject with hyperglycemia: Fasting blood glucose > 300 and/or with any of the above symptoms:

1. Contact a physician investigator to evaluate the subject. Physician investigator will make the clinical decision if the patient should have rapid-acting insulin administered and monitored, or referred to the nearest emergency department or can be safely discharged to their home.
2. The patient will not have OMT/OMT-sham treatment given at that specific research encounter

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type II diabetes
* Able to provide consent for participation
* Currently taking only oral diabetic medication(s)
* Prior hemoglobin A1C test result
* Able to fast for the glucose measurements
* Able to complete the intake and consent documents

Exclusion Criteria:

* Insulin dependent diabetes
* Unable or unwilling to provide informed consent
* Unable to fast for the glucose measurements
* Have an absolute contraindication to OMT (i.e. Acute fracture, joint dislocation, an open wound or infection)
* Pregnant women

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose | 3 months
  Short term fasting glucose levels

SECONDARY OUTCOMES:
A1C | 3 months
  Short term A1C levels

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Rivera-Martinez, DO, Principal Investigator — New York Institute of Technology
Locations (2):
- United States (2):
  - NYIT Family Health Care Center, Central Islip, New York
  - NYIT Academic Health Care Center - Riland Bldg., Old Westbury, New York

IPD SHARING:
Plan to Share IPD: Yes
The investigators will aim to present preliminary findings at poster presentation at American Academy of Osteopathy and American College of Osteopathic Family Medicine conferences and the final results at the American Osteopathic Association (AOA) OMED. The final results will be published in a peer review journal such as the Journal of the American Osteopathic Association or Endocrine Disorders. The authors would offer training of the Type II diabetes OMM treatment protocol utilized in this study as a training workshop at local and national conferences to enable other physicians who practice OMM to use it effectively. NYITCOM would assist in publicizing the research findings via the college's website and through our Public Relations/events coordinator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Six months after the completion of the study
Access Criteria: As determined by the publication journal

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Lindstrom J, Ilanne-Parikka P, Peltonen M, Aunola S, Eriksson JG, Hemio K, Hamalainen H, Harkonen P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Paturi M, Sundvall J, Valle TT, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Sustained reduction in the incidence of type 2 diabetes by lifestyle intervention: follow-up of the Finnish Diabetes Prevention Study. Lancet. 2006 Nov 11;368(9548):1673-9. doi: 10.1016/S0140-6736(06)69701-8. PMID 17098085
- [Background] Licciardone JC. Rediscovering the classic osteopathic literature to advance contemporary patient-oriented research: A new look at diabetes mellitus. Osteopath Med Prim Care. 2008 Jul 21;2:9. doi: 10.1186/1750-4732-2-9. PMID 18644129
- [Background] Shubrook JH Jr, Johnson AW. An osteopathic approach to type 2 diabetes mellitus. J Am Osteopath Assoc. 2011 Sep;111(9):531-7. PMID 21955532
- [Background] Johnson AW, Shubrook JH Jr. Role of osteopathic structural diagnosis and osteopathic manipulative treatment for diabetes mellitus and its complications. J Am Osteopath Assoc. 2013 Nov;113(11):829-36. doi: 10.7556/jaoa.2013.058. PMID 24174504
- [Background] Van Ravenswaay VJ, Hain SJ, Grasso S, Shubrook JH. Effects of Osteopathic Manipulative Treatment on Diabetic Gastroparesis. J Am Osteopath Assoc. 2015 Jul;115(7):452-8. doi: 10.7556/jaoa.2015.091. PMID 26111133
- [Background] Mendes GF, Nogueira JA, Reis CE, de Meiners MM, Dullius J. Diabetes education program with emphasis on physical exercise in subjects with type 2 diabetes: a community-based quasi-experimental study. J Sports Med Phys Fitness. 2017 Jun;57(6):850-858. doi: 10.23736/S0022-4707.16.06261-7. Epub 2016 May 24. PMID 27215770
- [Background] Licciardone JC, Fulda KG, Stoll ST, Gamber RG, Cage AC. A case-control study of osteopathic palpatory findings in type 2 diabetes mellitus. Osteopath Med Prim Care. 2007 Feb 8;1:6. doi: 10.1186/1750-4732-1-6. PMID 17371582